CLINICAL TRIAL: NCT03667235
Title: 10 Versus 20 Minutes Treatment of Human Pericardium With Glutaraldehyde in OZAKI Procedure
Acronym: 10vs20-OZAKI
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01334; ch17Reuthebuch2
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Aortic Valve Surgery
Keywords: OZAKI technique
MeSH Terms: interventions — Glutaral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Leftover tissues from the OZAKI procedure (excess of pericardium and calcified aortic valve leaflets) will be fixed in glutaraldehyde in the operation room and stored in sterile tubes in Phosphate Buffered Saline(PBS) and transferred at room temperature to the lab where it will be stored in a lab fridge at 4°C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment of human pericardium with glutaraldehyde in OZAKI procedure — 10 versus 20 minutes treatment of human pericardium with 0.6% glutaraldehyde in OZAKI procedure
Other: Treatment of human aortic valve tissue with glutaraldehyde — 10 versus 20 minutes treatment of human aortic valve tissue with 0.6%glutaraldehyde

SUMMARY:
To compare mechanic and thermic stability of pericardium fixated either with 0.6% glutaraldehyde for 10 minutes or with 0.6% glutaraldehyde for 20 minutes

DETAILED DESCRIPTION:
Autologous pericardium for aortic valve reconstruction is treated with 0.6% glutaraldehyde for 10 minutes to improve stability (OKAZI technique).

This study investigates whether treatment with 0.6% glutaraldehyde for 20 minutes improves mechanic and thermic stability of autologous pericardial tissue. Autologous pericardium remaining after aortic valve reconstruction surgery is used.

To investigate 10 versus 20 minutes treatment of removed original aortic valve tissue with glutaraldehyde as a reference.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing aortic valve surgery with sufficient leftover tissues from the OZAKI procedure (excess of pericardium and calcified aortic valve leaflets)

Exclusion Criteria:

* denial of consent
* insufficient leftover tissues from the OZAKI procedure
* patients after thoracic radiation or surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing aortic valve surgery with OZAKI technique at Universitätsspital Basel/ Switzerland
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
mechanic stability tests to investigate uniaxial and cyclical tensile properties | 4 days after surgery
  mechanical tests include the use of a universal test machine (MTS Bionix, Department of Bioengineering of Universitaetsspital Basel) for:
  * uniaxial ultimate tensile strength (UTS) test;
  * cyclical tensile stretching of the tissue in order to investigate its viscoelastic properties
thermic stability by using constant force at linearly increasing temperature | 4 days after surgery
  constant force at linearly increasing temperature: Thermal stability tests will be conducted on 20 x 4 mm stripes by the imposition of a constant load (approximately 1N) submerged in a saline-solution bath. The temperature of the bath will be increased at a rate of approximately 2.5-5 °C/min, and the sample cross-section will be measured by means of a high-resolution camera (Canon EOS, Japan)

SECONDARY OUTCOMES:
histologic analysis of collagen fiber organization and quantification | 4 days after surgery
  histologic analysis by Scanning Electrical Microscopy (SEM) and using Picrosirius staining to identify the types I and IV collagen
Pronase testing to analyse enzymatic degradation | 4 days after surgery
  Pronase testing to analyse enzymatic degradation

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, PD Dr. med, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland